CLINICAL TRIAL: NCT06595368
Title: A Randomized Controlled Trial Comparing the Efficacy of Vimala Massage Versus Hydrotherapy on Clinical Outcomes in Neonatal Hyperbilirubinemia
Brief Title: Comparing the Effect of Vimala Massage Versus Hydrotherapy on the Clinical Outcomes of Neonatal Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Wardany Abdelaal Mohamed, assistant professor of pediatric nursing, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KafrelsheikhU3
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Consisted of 30 newborns who will receive conventional hospital care with no additional interventions.
- Study group I (Vimala group) (Experimental): Consisted of 30 neonates who will receive Vimala massage.
  Interventions: Procedure: Vimala massage
- Study group II (Hydrotherapy) (Active Comparator): Consisted of 30 neonates who will receive hydrotherapy.
  Interventions: Procedure: Hydrotherapy

INTERVENTIONS:
Procedure: Vimala massage — The massage will be given three times per day, each lasting 15 minutes and planned one hour after the first feeding of each shift.
  Arms: Study group I (Vimala group)
Procedure: Hydrotherapy — Hydrotherapy will be applied two times per day before feeding, each lasting 5-10 min.
  Arms: Study group II (Hydrotherapy)

SUMMARY:
The aim of this study is to evaluate the effect of Vimala massage versus hydrotherapy on the clinical outcomes of neonatal hyperbilirubinemia.

DETAILED DESCRIPTION:
The researchers explained the study's aim, benefits, and procedures for participation, after that the parents of the neonates provided an informed consent. Neonatal baseline data was collected from their records on the first day of admission for the three groups prior to intervention in order to identify neonates who meet the required criteria of the study. then the participants were selected and divided randomly (using a simple random method) into three equal groups. One subject for the control group, one for the study group (I), then the other for study group (II), and so on, distributed the participants into three equivalent groups as fellow:

Control Group: Consisted of 30 newborns who will receive conventional hospital care with no additional interventions.

Study Group (I): Consisted of 30 neonates who will receive Vimala massage. The massage will be given three times per day, each lasting 15 minutes and planned one hour after the first feeding of each shift.

Study Group (II): Consisted of 30 neonates who will receive hydrotherapy. It will be applied two times per day before feeding, each lasting 5-10 min.

ELIGIBILITY:
Inclusion Criteria:

full-term neonates aged 37- 42 weeks of gestation with a birth weight of ≥1500 g and a five-minute Apgar score of seven or above. Furthermore, the newborn with physiological jaundice will be admitted for phototherapy from the first to the tenth day, and the infant's vital signs will remain normal

Exclusion Criteria:

* major congenital malformations, intestinal obstruction, congenital heart disease, sepsis, neonates with a disease that disrupts skin integrity (epidermolysis bullosa, ichthyosis, collodion baby).

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Total serum bilirubin level on Total serum bilirubin level monitoring sheet | Daily measurement from first day of neonate's admission to day 5 of admission
  Total serum bilirubin level monitoring sheet: it includes 2 tests of total serum bilirubin level & indirect serum bilirubin tests. The daily measurement will be done, its primary purpose is to evaluate the effect of Vimala massage and hydrotherapy on newborns with Jaundice undergoing phototherapy. Bilirubin will be measured using microassay.
Change from baseline of neonate's weight on Bilirubin excretion monitoring sheet | Daily measurement from first day of neonate's admission to day 5 of admission
  Bilirubin excretion monitoring sheet: it includes daily measurement of the neonate's weight
Change from baseline of neonate's number of diaper exchange to monitor the frequency of defection and amount of stool on Bilirubin excretion monitoring sheet | Daily measurement from first day of neonate's admission to day 5 of admission
  Bilirubin excretion monitoring sheet: it includes daily monitoring of infant's diaper exchange to monitor the frequency of defection and amount of stool
Change from baseline of neonate's total feeding amount on Bilirubin excretion monitoring sheet | Daily measurement from first day of neonate's admission to day 5 of admission
  Bilirubin excretion monitoring sheet: it includes daily monitoring of neonate's total feeding amount

SECONDARY OUTCOMES:
Estimate the time of jaundice regression and duration of phototherapy on Clinical efficacy monitoring tool | through 5 days from admission
  Clinical efficacy monitoring tool was developed by researchers after a review of relevant literature to assess the effectiveness of Vimala massage and Hydrotherapy in accelerating the regression time of jaundice.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No